CLINICAL TRIAL: NCT06107387
Title: Binge Eating Self-help for Teens (BEST): A Pilot and Feasibility Test of an Online Behavioral Intervention for Adolescents With Binge Eating and Elevated Weight
Brief Title: Binge Eating Self-help for Teens ONLINE Pilot and Feasibility Study
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000033103; 000 (Other: CTGTY)
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Binge Eating; Binge-Eating Disorder; Overweight or Obesity
MeSH Terms: conditions — Bulimia; Binge-Eating Disorder; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Binge Eating Self-help for Teens (Experimental): Participants will have 16 guided self-help sessions (4 months; weekly sessions for adolescents with parents joining monthly). Participants will complete daily self-monitoring of eating behaviors (timing of meals and snacks; whether or not a binge occurred) throughout treatment. Treatment sessions involve a self-help component, which includes brief videos that participants watch at home. Treatment sessions also involve a guidance component (brief consultation), which is 15-30 minutes on a secure videoconferencing platform (e.g., Zoom) between the therapist and the participant. These sessions focus on clarifying material, reviewing self-monitoring and looking for patterns, and problem-solving maladaptive thinking patterns and binge behaviors.
  Interventions: Behavioral: Binge Eating Self-help for Teens

INTERVENTIONS:
Behavioral: Binge Eating Self-help for Teens — Guided self-help intervention
  Other Names: BEST

SUMMARY:
This study is a pilot clinical trial of a new guided self-help CBT for binge eating. Participants will complete an intake assessment; following determination of eligibility, participants will then complete four months of treatment (weekly guided self-help sessions). At the end of treatment, participants will complete an interview with a research clinician to assess outcomes.

ELIGIBILITY:
Inclusion Criteria: To be included, adolescents must:

1. Be in the age range ≥12 years old and ≤17 years old;
2. Have a BMI that places them above the 85th percentile based on their age and sex;
3. Report 2 episodes of binge/LOC eating (feeling a loss of control while eating) per month for the past 3 months;
4. Be otherwise-healthy youth (i.e., no uncontrolled or serious medical conditions);
5. Read, comprehend, and write English at a sufficient level to complete study-related materials;
6. Provide a signed and dated written assent prior to study participation;
7. Provide a signed and dated written consent from one parent prior to study participant; and
8. Be available for participation in the study for 4 months.

Exclusion Criteria: Prospective participants will be excluded if the adolescent:

1. Has a medical or psychiatric condition that would require hospitalization or intensive care (e.g., neurological disorder, psychotic disorders, suicidality);
2. Has a medical or psychiatric condition that would prohibit them from engaging in behavioral treatment or moderate physical activity (e.g., cardiovascular problems);
3. Has uncontrolled medical condition(s) (e.g., uncontrolled diabetes or hypertension);
4. Is pregnant or breastfeeding;
5. Is taking medication(s) or participating in treatment(s) that could influence weight or appetite;
6. Began taking hormonal contraceptives less than 3 months prior;
7. Has a developmental or cognitive disorder (e.g., autism spectrum disorder);
8. Has a concurrent feeding/eating disorder (e.g., bulimia nervosa); or
9. Is participating in another clinical research study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Attendance | 4 months
  Number of participants attending >75% of sessions
Retention | 4 months
  Number of participants who attend through the end of treatment

SECONDARY OUTCOMES:
Treatment Credibility | 1 week
  Adolescent/parent treatment credibility (moderate or higher, study-specific face-valid treatment credibility form)
Treatment Satisfaction | 4 months
  Adolescent/parent/clinician treatment satisfaction (acceptable or higher, Client Satisfaction Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Janet A Lydecker, PhD, Principal Investigator — Yale University
Locations (1):
- Yale, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study. We are prioritizing individuals' privacy because they are children and binge eating and weight can be stigmatizing. We will consider requests to share individual-level data from other researchers if they are consistent with privacy protections.